CLINICAL TRIAL: NCT03688932
Title: Effects of Whole Body Vibration Associated With the Inspiratory Muscle Training Program on Functional Capacity, Balance and Muscle Metabolism
Brief Title: Effects of WBV Associated With IMT on Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helga Cecília Muniz de Souza, Msc, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WBV on Functionality
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Frail Elderly Syndrome
Keywords: aging; functional capacity; muscle metabolism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WBV + IMT (Experimental): Whole body vibration training associated with respiratory muscle training (WBV + IMT)
  Interventions: Other: WBV + IMT
- WBV + IMTsham (Active Comparator): Whole body vibration training associated with respiratory muscle training sham (WBV + IMTsham)
  Interventions: Other: WBV + IMTsham
- WBVsham + IMTsham (Sham Comparator): Whole body vibration training sham associated with respiratory muscle training sham (WBVsham + IMTsham)
  Interventions: Other: WBVsham + IMTsham

INTERVENTIONS:
Other: WBV + IMT — The whole body vibration training will be performed through a vibrating platform with three axes and vibration frequency set at 35 Hz. The amplitude used will be 02 to 04 mm.The inspiratory muscle training will be performed through a device that provides inspiratory resistance.
  Arms: WBV + IMT
Other: WBV + IMTsham — The whole body vibration training will be performed through a vibrating platform with three axes and vibration frequency set at 35 Hz. The amplitude used will be 02 to 04 mm.The inspiratory muscle training sham will be performed through a device without inspiratory resistance.
  Arms: WBV + IMTsham
Other: WBVsham + IMTsham — Whole body vibration training will be performed through a vibrating platform coupled to a device that generates non-therapeutic low frequency vibration. The simulation of inspiratory muscle training will be performed through a device with no inspiratory resistance.
  Arms: WBVsham + IMTsham

SUMMARY:
The pre-frail elderly are a population more vulnerable to diminished functionality and future disabilities. Thus, interventions focused on the prevention of sarcopenia are indicated to prevent dysfunction in this population. This study aims to evaluate the effects of whole body vibration training associated with inspiratory muscle training on functional outcomes, balance and muscle metabolism in pre-frail elderly women.

ELIGIBILITY:
Inclusion Criteria:

* To able to walk without assistance
* Good understanding to carry out the proposed tests, evaluated through the Mini Mental State Examination (MMSE).

Exclusion Criteria:

* Contraindication or difficulty to perform evaluation procedures
* Users of medications that interfere with the cardiovascular and / or muscular system
* Smokers
* Neuromuscular or degenerative diseases
* Pulmonary comorbidities
* Heart diseases and labyrinthitis

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Walking Distance | Change from Baseline walking distance at 3 months
  The walking distance will be assessed through the six-minute walk test.

SECONDARY OUTCOMES:
Balance | Change from Baseline balance at 3 months
  Static balance and dynamic balance will be evaluated through the Tinetti test
Functionality | Change from Baseline functionality at 3 months
  It will be evaluated through the Timed Up and Go (TUG) test.
Hand grip strength | Change from Baseline hand grip strength at 3 months
  The strength of the dominant hand will be evaluated by dynamometry.
Muscle Metabolism | Change from Baseline muscle metabolism at 3 months
  It will be assessed through the blood lactate and glucose rate after moderate physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil